CLINICAL TRIAL: NCT04035200
Title: A Phase 2, Randomized, Double-Blind, Multi-Center, Placebo-Controlled, Parallel-Group Study to Evaluate the Safety, Tolerability, and Efficacy of V117957 in Subjects With an Alcohol Use Disorder Who Are Experiencing Insomnia Associated With Alcohol Cessation
Brief Title: Safety, Tolerability and Efficacy Study of V117957 in Subjects With Insomnia Associated With Alcohol Cessation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imbrium Therapeutics (Industry)
Collaborators: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OAG2002
Record Dates: First submitted 2019-07-25; First posted 2019-07-29 (Actual); Results first posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- V117957 1 mg (Experimental): V117957 tablets taken orally at bedtime
  Interventions: Drug: V117957 tablets
- V117957 2 mg (Experimental): V117957 tablets taken orally at bedtime
  Interventions: Drug: V117957 tablets
- Placebo (Placebo Comparator): Placebo to match V117957 tablets taken orally at bedtime
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: V117957 tablets — V117957 tablets taken orally at bedtime
  Arms: V117957 1 mg; V117957 2 mg
Drug: Placebo — Tablets to match V117957
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and efficacy of V117957 in subjects with alcohol use disorder (AUD) who experience insomnia associated with alcohol cessation, compared to placebo.

ELIGIBILITY:
Key Inclusion Criteria include:

* Male or female, 18-64 years of age with a body weight of 50-100 kg (110-220 lbs) and a body mass index (BMI) of 18-32 kg/m2.
* Otherwise healthy as determined by medical evaluation that includes: medical history, physical examination, neurological exam, laboratory tests, vital signs, and cardiac monitoring.
* History of moderate or severe alcohol use disorder (AUD) categorized based on Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM-5) criteria, as follows:

  * Moderate as defined by presence of 4-5 of the 11 criteria
  * Severe as defined by the presence of ≥ 6 of the 11 criteria.
* At least 3 weeks and not more than 6 months since last alcoholic beverage intake at the time of study screening. Any subject who completed an alcohol detoxification program must be at least 7 days from completion of the program at the time of screening.
* Persistent insomnia that emerged or worsened during AUD period, or during or after alcohol cessation characterized by a study-specific sleep diary.
* A female participant is eligible to participate if she is not pregnant and not breastfeeding. Both females of childbearing potential and nonsurgically sterilized males with a sexual partner of childbearing potential must be willing to use adequate and reliable contraception throughout the study.
* Willing to refrain from a behavioral or other treatment program for insomnia during participation in the study.

Key Exclusion Criteria include:

* Current diagnosis of a sleep-related breathing disorder including obstructive sleep apnea (with or without continuous positive airway pressure (CPAP) treatment), periodic limb movement disorder, restless legs syndrome, circadian rhythm sleep disorder or narcolepsy.
* An apnea-hypopnea index (AHI) score of >10 or a periodic limb movement arousal index (PLMAI) score of > 15 recorded during the screening period PSG.
* Documented history of insomnia prior to onset of the alcohol use disorder (AUD), which did not worsen during the AUD period or during or after alcohol cessation.
* Comorbid conditions which interfere with normal sleep pattern or the evaluation of next day residual effects.
* Any lifetime history of suicidal ideation or behavior.
* History of or any current conditions that might interfere with drug absorption, distribution, metabolism, or excretion (including any surgical interventions for weight loss).
* Any history of seizures (except related to alcohol withdrawal) or head trauma with sequelae.
* Known history of testing positive for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV).
* History of diagnosed, active liver disease or elevated liver enzymes/bilirubin.
* History of kidney stones or renal insufficiency or abnormal kidney function at screening.
* Uncontrolled hypertension (> 140 mm Hg systolic / 90 mm Hg diastolic).
* Use of any medication that affects sleep and/or wake function during the week before starting the screening period.
* Subjects currently undergoing treatment of other addictions in addition to alcohol.
* Excessive caffeine consumption.
* Positive urine drug screen for prohibited substances, except for cannabis on a case-by-case basis.
* History of drug use disorder over the past year, other than alcohol/nicotine/caffeine/cannabis.
* Plans to travel across more than 3 time zones in the 2 weeks before screening, or during study participation.
* Night or rotating shift worker.
* Any history and/or current evidence of other medical (eg, cardiac, respiratory, gastrointestinal, renal, malignancy other than basal cell carcinoma), neurological, or psychiatric conditions that, in the opinion of the investigator, could affect the subject's safety or interfere with the study.

Other protocol-specific inclusion/exclusion criteria may apply.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - California Clinical Trials Medical Group, Glendale, California
  - Artemis Institute for Clinical Research, Riverside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - CITrials, Santa Ana, California
  - SDS Clinical Trials, Inc., Santa Ana, California
  - St. Francis Medical Institute, Clearwater, Florida
  - Research Centers of America, Hollywood, Florida
  - Research Centers of America, LLC, Miami, Florida
  - Innovative Clinical Research, Inc., Miami Lakes, Florida
  - NeuroTrials Research Inc, Atlanta, Georgia
  - Investigational Site, Chevy Chase, Maryland
  - Sleep Disorders Centers of the Mid Atlantic, Glen Burnie, Maryland
  - Wake Research - Clinical Research Center of Nevada, LLC, Las Vegas, Nevada
  - SPRI Clinical Trials, Brooklyn, New York
  - Clinilabs Drug Development Corporation, New York, New York
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Advanced Medical Trials, Georgetown, Texas

REFERENCES:
- [Derived] Whiteside GT, Kyle DJ, Kapil RP, Cipriano A, He E, Zhou M, Shet MS, Hummel M, Knappenberger T, Fukumura K, Matsuo Y, Uehira M, Hiroyama S, Takai N, Willsie SK, Harris SC. The nociceptin/orphanin FQ receptor partial agonist sunobinop promotes non-REM sleep in rodents and patients with insomnia. J Clin Invest. 2024 Jan 2;134(1):e171172. doi: 10.1172/JCI171172. PMID 37883189

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multi-center study conducted at study sites in the US.
Period: Overall Study
Arm/Group | V117957 1 mg | V117957 2 mg | Placebo
Started | 38 | 38 | 38
Completed | 36 | 31 | 34
Not Completed | 2 | 7 | 4
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 4 | 4
Not completed — COVID-19 | 1 | 0 | 0
Not completed — Early Termination | 0 | 1 | 0
Not completed — Non-compliance | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V117957 1 mg | V117957 2 mg | Placebo | Total
Number analyzed (Participants) | 38 | 38 | 38 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (12.85) | 45.2 (13.01) | 44.9 (12.18) | 44.5 (12.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 16 | 24 | 61
  Male | 17 | 22 | 14 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 11 | 6 | 23
  White | 31 | 26 | 32 | 89
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Wakefulness After Sleep Onset (WASO) Measured by Polysomnography (PSG)
Description: Wakefulness After Sleep Onset, as measured by PSG, was defined as wake time after persistent sleep (wake time during sleep plus wake time after sleep, expressed in minutes). Nights 1 / 2 is the average of the PSG measurements taken during the first two nights of study drug exposure. Nights 20 / 21 is the average of the PSG measurements taken during nights 20 and 21 of study drug exposure.
Time Frame: Baseline, Nights 1 / 2, Nights 20 / 21
Population: Full analysis population: The group of subjects who were randomly assigned to 1 of the 3 treatment groups, received study drug, and had at least 1 valid postdose efficacy measurement.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | V117957 1 mg | V117957 2 mg | Placebo
Number analyzed (Participants) | 38 | 37 | 38
Minutes
  Baseline | 100.88 (45.098) | 99.70 (36.496) | 103.51 (32.456)
  Nights 1 / 2 | 48.64 (28.453) | 42.44 (28.189) | 63.00 (29.349)
  Nights 20 / 21: number analyzed (Participants) | 36 | 31 | 32
  Nights 20 / 21 | 50.56 (34.115) | 46.17 (27.275) | 64.43 (33.999)

2. Secondary Outcome: Change From Baseline in Mean Sleep Efficiency (SE)
Description: Sleep efficiency, as measured by PSG, is defined as Total Sleep Time (TST), divided by total recording time, multiplied by 100.
  Nights 1 / 2 is the average of the PSG measurements taken during the first two nights of study drug exposure. Nights 20 / 21 is the average of the PSG measurements taken during nights 20 and 21 of study drug exposure.
Time Frame: Baseline, Nights 1 / 2, Nights 20 / 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | V117957 1 mg | V117957 2 mg | Placebo
Number analyzed (Participants) | 38 | 37 | 38
Percent
  Baseline | 64.54 (11.502) | 67.18 (9.919) | 63.17 (12.825)
  Nights 1 / 2 | 82.00 (10.810) | 85.55 (7.953) | 77.64 (9.950)
  Nights 20 / 21: number analyzed (Participants) | 36 | 31 | 32
  Nights 20 / 21 | 79.46 (10.516) | 84.89 (7.456) | 78.38 (8.890)

3. Secondary Outcome: Change From Baseline in Mean Latency to Persistent Sleep (LPS)
Description: Latency to onset of persistent sleep (LPS), as measured by PSG, is defined as time from lights-off to the first of 20 consecutive periods of non-wake sleep stages. Latency to persistent sleep is reported in minutes.
  Nights 1 / 2 is the average of the PSG measurements taken during the first two nights of study drug exposure. Nights 20 / 21 is the average of the PSG measurements taken during nights 20 and 21 of study drug exposure.
Time Frame: Baseline, Nights 1 / 2, Nights 20 / 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | V117957 1 mg | V117957 2 mg | Placebo
Number analyzed (Participants) | 38 | 37 | 38
Minutes
  Baseline | 76.63 (34.305) | 66.30 (25.653) | 81.58 (48.928)
  Nights 1 / 2 | 43.03 (38.542) | 31.31 (20.593) | 51.74 (37.243)
  Nights 20 / 21: number analyzed (Participants) | 36 | 31 | 32
  Nights 20 / 21 | 53.48 (47.123) | 31.70 (25.709) | 47.42 (31.165)

4. Secondary Outcome: Change From Baseline in Mean Total Sleep Time (TST)
Description: Total sleep time, as measured by PSG, is the duration of rapid eye movement (REM) plus NREM (stages N1 + N2 + N3) during time in bed.
  Nights 1 / 2 is the average of the PSG measurements taken during the first two nights of study drug exposure. Nights 20 / 21 is the average of the PSG measurements taken during nights 20 and 21 of study drug exposure.
Time Frame: Baseline, Nights 1 / 2, Nights 20 / 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | V117957 1 mg | V117957 2 mg | Placebo
Number analyzed (Participants) | 38 | 37 | 38
Minutes
  Baseline | 309.87 (55.265) | 323.11 (48.065) | 303.24 (61.559)
  Nights 1 / 2 | 393.80 (51.677) | 410.12 (38.771) | 372.68 (47.771)
  Nights 20 / 21: number analyzed (Participants) | 36 | 31 | 32
  Nights 20 / 21 | 381.65 (50.528) | 407.45 (35.765) | 376.26 (42.640)

5. Secondary Outcome: Change From Baseline in Mean Number of Awakenings (NAW)
Description: Sleep component as measured by PSG. Number of awakenings is determined from persistent sleep to lights-on. An awakening is defined as a PSG recording of at least 2 consecutive wake periods.
  Nights 1 / 2 is the average of the PSG measurements taken during the first two nights of study drug exposure. Nights 20 / 21 is the average of the PSG measurements taken during nights 20 and 21 of study drug exposure.
Time Frame: Baseline, Nights 1 / 2, Nights 20 / 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of Awakenings
Arm/Group | V117957 1 mg | V117957 2 mg | Placebo
Number analyzed (Participants) | 38 | 37 | 38
Number of Awakenings
  Baseline | 10.70 (5.733) | 14.05 (5.101) | 10.32 (5.609)
  Nights 1 / 2 | 8.25 (3.860) | 9.62 (5.599) | 10.20 (4.256)
  Nights 20 / 21: number analyzed (Participants) | 36 | 31 | 32
  Nights 20 / 21 | 9.29 (5.114) | 10.63 (6.055) | 10.28 (5.575)

6. Secondary Outcome: Change From Baseline in Subjective Sleep Quality (sSleep)
Description: Self-reported sleep outcome measured by subject diary data. Scores have a range of 1 to 5, with 1 being equal to "Very Poor" and 5 being equal to "'Very Good."
  Nights 1 / 2 is the average of the measurements taken during the first two nights of study drug exposure. Nights 20 / 21 is the average of the measurements taken during nights 20 and 21 of study drug exposure.
Time Frame: Baseline, Nights 1 / 2, Nights 20 / 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | V117957 1 mg | V117957 2 mg | Placebo
Number analyzed (Participants) | 38 | 37 | 38
score on a scale
  Baseline: number analyzed (Participants) | 35 | 30 | 33
  Baseline | 1.80 (0.686) | 1.82 (0.683) | 1.99 (0.727)
  Nights 1 / 2: number analyzed (Participants) | 38 | 36 | 38
  Nights 1 / 2 | 2.72 (0.984) | 2.92 (1.004) | 2.64 (0.734)
  Nights 20 / 21: number analyzed (Participants) | 36 | 34 | 35
  Nights 20 / 21 | 2.94 (0.989) | 3.11 (1.027) | 3.20 (0.841)

7. Secondary Outcome: Change From Baseline in Subjective Total Sleep Time (sTST)
Description: Self-reported sleep outcome measured by subject diary data. Total sleep time is reported in minutes.
  Nights 1 / 2 is the average of the measurements taken during the first two nights of study drug exposure. Nights 20 / 21 is the average of the measurements taken during nights 20 and 21 of study drug exposure.
Time Frame: Baseline, Nights 1 / 2, Nights 20 / 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | V117957 1 mg | V117957 2 mg | Placebo
Number analyzed (Participants) | 38 | 37 | 38
Minutes
  Baseline: number analyzed (Participants) | 35 | 30 | 33
  Baseline | 296.42 (45.586) | 304.60 (50.458) | 315.05 (56.092)
  Nights 1 / 2: number analyzed (Participants) | 38 | 36 | 38
  Nights 1 / 2 | 355.82 (69.903) | 357.35 (80.198) | 350.64 (51.843)
  Nights 20 / 21: number analyzed (Participants) | 36 | 34 | 35
  Nights 20 / 21 | 366.14 (59.562) | 385.13 (71.181) | 384.13 (58.830)

8. Secondary Outcome: Change From Baseline in Subjective Wakefulness After Sleep Onset (sWASO)
Description: Self-reported sleep outcome measured by subject diary data. WASO is defined as wake time after persistent sleep (wake time during sleep plus wake time after sleep, expressed in minutes).
  Nights 1 / 2 is the average of the measurements taken during the first two nights of study drug exposure. Nights 20 / 21 is the average of the measurements taken during nights 20 and 21 of study drug exposure.
Time Frame: Baseline, Nights 1 / 2, Nights 20 / 21
Population: \Full analysis population: The group of subjects who were randomly assigned to 1 of the 3 treatment groups, received study drug, and had at least 1 valid postdose efficacy measurement.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | V117957 1 mg | V117957 2 mg | Placebo
Number analyzed (Participants) | 38 | 37 | 38
Minutes
  Baseline: number analyzed (Participants) | 35 | 30 | 33
  Baseline | 92.51 (42.137) | 85.93 (42.222) | 83.49 (63.929)
  Nights 1 / 2: number analyzed (Participants) | 36 | 33 | 38
  Nights 1 / 2 | 63.77 (63.476) | 59.48 (55.546) | 55.72 (34.974)
  Nights 20 / 21: number analyzed (Participants) | 36 | 31 | 35
  Nights 20 / 21 | 51.53 (40.574) | 54.21 (44.666) | 46.84 (32.499)

9. Secondary Outcome: Change From Baseline in Subjective Sleep Onset Latency (sSOL)
Description: Self-reported sleep outcome measured by subject diary data. Sleep onset latency (SOL) is the time it takes to fall asleep after turning the lights out.
  Nights 1 / 2 is the average of the measurements taken during the first two nights of study drug exposure. Nights 20 / 21 is the average of the measurements taken during nights 20 and 21 of study drug exposure.
Time Frame: Baseline, Nights 1 / 2, Nights 20 / 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | V117957 1 mg | V117957 2 mg | Placebo
Number analyzed (Participants) | 38 | 37 | 38
Minutes
  Baseline: number analyzed (Participants) | 35 | 30 | 33
  Baseline | 74.54 (30.022) | 75.84 (31.274) | 63.45 (19.795)
  Nights 1 / 2: number analyzed (Participants) | 38 | 36 | 38
  Nights 1 / 2 | 54.42 (29.031) | 50.53 (32.579) | 57.24 (28.375)
  Nights 20 / 21: number analyzed (Participants) | 36 | 34 | 35
  Nights 20 / 21 | 63.13 (32.740) | 47.14 (24.289) | 47.68 (33.170)

10. Secondary Outcome: Change From Baseline in Subjective Sleep Efficiency (sSE)
Description: Self-reported sleep outcome measured by subject diary data. Sleep efficiency (SE) is calculated by dividing the time asleep by the total time in bed multiplied by 100 (SE is reported as percent).
  Nights 1 / 2 is the average of the measurements taken during the first two nights of study drug exposure. Nights 20 / 21 is the average of the measurements taken during nights 20 and 21 of study drug exposure.
Time Frame: Baseline, Nights 1 / 2, Nights 20 / 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | V117957 1 mg | V117957 2 mg | Placebo
Number analyzed (Participants) | 38 | 37 | 38
Percent
  Baseline: number analyzed (Participants) | 26 | 23 | 25
  Baseline | 61.51 (8.768) | 63.14 (8.898) | 63.50 (10.924)
  Nights 1 / 2: number analyzed (Participants) | 38 | 36 | 38
  Nights 1 / 2 | 73.26 (14.436) | 73.72 (16.661) | 71.53 (10.229)
  Nights 20 / 21: number analyzed (Participants) | 36 | 34 | 35
  Nights 20 / 21 | 73.74 (11.925) | 76.78 (12.383) | 75.88 (11.743)

11. Secondary Outcome: Change From Baseline in Subjective Number of Awakenings (sNAW)
Description: Self-reported sleep outcome measured by subject diary data. The subject recorded the number of awakenings in the diary.
  Nights 1 / 2 is the average of the measurements taken during the first two nights of study drug exposure. Nights 20 / 21 is the average of the measurements taken during nights 20 and 21 of study drug exposure.
Time Frame: Baseline, Nights 1 / 2, Nights 20 / 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of Awakenings
Arm/Group | V117957 1 mg | V117957 2 mg | Placebo
Number analyzed (Participants) | 38 | 37 | 38
Number of Awakenings
  Baseline: number analyzed (Participants) | 35 | 30 | 33
  Baseline | 2.49 (1.100) | 2.24 (1.013) | 2.37 (0.984)
  Nights 1 / 2: number analyzed (Participants) | 38 | 36 | 38
  Nights 1 / 2 | 1.87 (1.245) | 2.14 (2.703) | 2.63 (1.647)
  Nights 20 / 21: number analyzed (Participants) | 36 | 34 | 35
  Nights 20 / 21 | 1.42 (1.049) | 1.30 (0.815) | 1.66 (1.405)

12. Secondary Outcome: Change From Baseline in Subjective Morning Sleepiness on Awakening
Description: Self-reported sleep outcome measured by subject diary data. Individual scores have a range of 1 to 5, with 1 being equal to "Not at All Rested" and 5 being equal to "Very Well Rested." Nights 1 / 2 is the average of the measurements taken during the first two nights of study drug exposure. Nights 20 / 21 is the average of the measurements taken during nights 20 and 21 of study drug exposure.
Time Frame: Baseline, Nights 1 / 2, Nights 20 / 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | V117957 1 mg | V117957 2 mg | Placebo
Number analyzed (Participants) | 38 | 37 | 38
score on a scale
  Baseline: number analyzed (Participants) | 35 | 30 | 33
  Baseline | 1.54 (0.655) | 1.60 (0.613) | 1.72 (0.611)
  Nights 1 /2: number analyzed (Participants) | 38 | 36 | 38
  Nights 1 /2 | 2.23 (0.870) | 2.19 (0.847) | 2.24 (0.695)
  Nights 20 / 21: number analyzed (Participants) | 36 | 34 | 35
  Nights 20 / 21 | 2.52 (0.979) | 2.69 (1.158) | 2.81 (0.937)

13. Secondary Outcome: Proportion of Responders to V117957 1 mg and 2 mg Compared to Placebo
Description: The proportion of responders is based on subjects meeting or exceeding WASO (wakefulness after sleep onset) 15 minute threshold as derived from polysomnography (PSG).
  Nights 1 / 2 is the average of the measurements taken during the first two nights of study drug exposure. Nights 20 / 21 is the average of the measurements taken during nights 20 and 21 of study drug exposure.
Time Frame: Nights 1 / 2, Nights 20 / 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | V117957 1 mg | V117957 2 mg | Placebo
Number analyzed (Participants) | 38 | 37 | 38
Participants
  Responder - Nights 1 / 2 - Threshold 15 minutes | 29 | 33 | 30
  Responder - Nights 20 / 21 - Threshold 15 minutes: number analyzed (Participants) | 36 | 31 | 32
  Responder - Nights 20 / 21 - Threshold 15 minutes | 33 | 27 | 25

14. Secondary Outcome: Occurrence of Rebound Insomnia During the Washout/Follow-up Period
Description: Rebound insomnia is defined as a worsening of sleep compared with pretreatment. The comparison is based on the Wakefulness After Sleep Onset (WASO) measured by PSG of the Washout/Follow-up Period versus Baseline. If the LS means for WASO for the Washout/Follow-up Period is lower than Baseline, then no rebound insomnia was suggested. Nights 22 / 23 is the average of the measurements taken during nights 22 and 23 (Washout Period).
Time Frame: Baseline Compared to Washout/Follow-up Period (Nights 22 / 23)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | V117957 1 mg | V117957 2 mg | Placebo
Number analyzed (Participants) | 38 | 37 | 38
Minutes
  Baseline | 100.88 (45.098) | 99.70 (36.496) | 103.51 (32.456)
  Washout/Follow-up Period: number analyzed (Participants) | 36 | 30 | 32
  Washout/Follow-up Period | 78.82 (48.048) | 94.23 (58.961) | 65.03 (33.942)

15. Secondary Outcome: Next Day Residual Effects as Determined by Digit Symbol Substitution Test (DSST).
Description: The DSST explores attention and psychomotor speed by measuring total correct responses. The maximum score is 165. Higher scores represent better outcome/improvement.
Time Frame: Baseline, Night 2, Night 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Correct Responses
Arm/Group | V117957 1 mg | V117957 2 mg | Placebo
Number analyzed (Participants) | 38 | 37 | 38
Correct Responses
  Baseline - Total correct responses | 49.0 (17.82) | 46.4 (15.85) | 46.2 (18.95)
  Night 2;10-hours postdose - Total correct responses: number analyzed (Participants) | 36 | 35 | 38
  Night 2;10-hours postdose - Total correct responses | 51.6 (16.06) | 51.7 (13.83) | 54.8 (13.58)
  Night 21; 10-hours postdose - Total correct responses: number analyzed (Participants) | 35 | 31 | 32
  Night 21; 10-hours postdose - Total correct responses | 52.0 (16.67) | 52.6 (18.65) | 54.3 (15.66)

16. Secondary Outcome: Next Day Residual Effects as Determined by Karolinska Sleepiness Scale (KSS)
Description: The KSS is a 9-point Likert scale (range: 1 = "extremely alert" to 9 = "very sleepy") that measures level of sleepiness.
Time Frame: Baseline, Night 2 (9- and 10-hours postdose), Night 21 (9- and 10-hours postdose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | V117957 1 mg | V117957 2 mg | Placebo
Number analyzed (Participants) | 34 | 32 | 32
score on a scale
  Baseline | 4.3 (2.30) | 4.4 (2.23) | 4.4 (2.09)
  Night 2 - 9 hours postdose: number analyzed (Participants) | 32 | 27 | 31
  Night 2 - 9 hours postdose | 4.2 (1.94) | 4.7 (2.17) | 4.3 (2.06)
  Night 2 - 10 hours postdose: number analyzed (Participants) | 30 | 27 | 31
  Night 2 - 10 hours postdose | 3.8 (1.94) | 4.0 (2.03) | 3.9 (1.93)
  Night 21 - 9 hours postdose: number analyzed (Participants) | 28 | 24 | 27
  Night 21 - 9 hours postdose | 4.1 (1.99) | 4.5 (2.34) | 3.9 (1.75)
  Night 21 - 10 hours postdose: number analyzed (Participants) | 28 | 24 | 27
  Night 21 - 10 hours postdose | 3.8 (2.02) | 4.0 (1.88) | 3.1 (1.31)

17. Secondary Outcome: Next Day Residual Effects as Determined by Profile of Mood States (POMS) - Brief
Description: The POMS-Brief contains 30 questions that assess mood states. Scores for each question range 0 = not at all to 4 = extremely. Total mood disturbance assessment is the total of the subject's subscales scores on anger/hostility, confusion/bewilderment, depression/dejection, fatigue/inertia, tension/anxiety, and vigor/activity. Total scores range from 0-120 and a higher total score indicates more mood disturbance.
Time Frame: Baseline, Night 2, Night 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | V117957 1 mg | V117957 2 mg | Placebo
Number analyzed (Participants) | 38 | 37 | 38
score on a scale
  Baseline: number analyzed (Participants) | 35 | 32 | 32
  Baseline | 13.54 (23.612) | 12.03 (15.658) | 11.80 (16.863)
  Night 2: number analyzed (Participants) | 31 | 28 | 32
  Night 2 | 5.41 (16.732) | 5.46 (14.674) | 6.34 (15.905)
  Night 21: number analyzed (Participants) | 29 | 24 | 26
  Night 21 | 2.02 (15.075) | 5.22 (13.630) | 1.58 (16.305)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported from the start of study participation up to 3 weeks. All-cause mortality and serious adverse events were reported from the start of study participation up to 30 days after last study drug dose (approximately 7 weeks).
Arm/Group | V117957 1 mg | V117957 2 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 5/38 | 14/38 | 7/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | V117957 1 mg (N=38) | V117957 2 mg (N=38) | Placebo (N=38)
Somnolence (Nervous system disorders) | 2 | 10 | 0
Headache (Nervous system disorders) | 3 | 1 | 2
Nausea (Gastrointestinal disorders) | 2 | 1 | 3
Fatigue (General disorders) | 0 | 2 | 2
Blood triglycerides increased (Investigations) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-27): https://cdn.clinicaltrials.gov/large-docs/00/NCT04035200/Prot_SAP_000.pdf